CLINICAL TRIAL: NCT04520009
Title: Randomize Everyone: Creating Valid Instrumental Variables for Learning Health Care Systems
Brief Title: EHR Embedded Comparative Effectiveness Studies--CPS
Acronym: EHR-CPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Trustees of Dartmouth College (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Tor D. Tosteson, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SFD20160
Record Dates: First submitted 2020-01-10; First posted 2020-08-20 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: Disk Herniated Lumbar
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity Restriction (Active Comparator): Discharge orders for activity restriction
  Interventions: Behavioral: Activity Restriction
- Activity As Tolerated (Active Comparator): Discharge orders written for activity as tolerated
  Interventions: Behavioral: Activity as Tolerated

INTERVENTIONS:
Behavioral: Activity Restriction — Standard post-operative activity instructions (i.e., no bending, twisting, or lifting more than 10 lbs for 4 weeks, no return to work until cleared to do so).
  Arms: Activity Restriction
Behavioral: Activity as Tolerated — Instructions advising activity as tolerated and return to work based on patient discretion
  Arms: Activity As Tolerated

SUMMARY:
Randomize Everyone is a research project to develop new informatics systems and statistical methods for supporting randomization processes in EHR systems to do comparative effectiveness research. Two demonstration projects are being conducted in the Dartmouth Hitchcock Medical Center, designed to evaluate different weight loss interventions and common practices in the treatment of chronic low back pain.

DETAILED DESCRIPTION:
EHR Embedded Comparative Effectiveness Studies-CPS will be held in the Center for Pain and Spine at Dartmouth-Hitchcock Medical Center. This study consists of randomizing enrollees to either activity restriction or no activity restriction following lumbar discectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18) able to consent
* Sufficient fluency in English
* Indications for discectomy
* Able to restrict activities or to resume activities as tolerated

Exclusion Criteria:

* Pregnant women
* Prisoners
* Children (<18).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor Tosteson, ScD, Principal Investigator — Dartmouth
Locations (1):
- Dartmouth-HItchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
No plans at this time share IPD

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Activity Restriction | Activity As Tolerated
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Activity Restriction | Activity As Tolerated | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (13.2) | 46.8 (17.2) | 46.5 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Compliance Rate With Assigned Treatment
Description: Compliance with assigned treatment as measured by presence of appropriate surgical discharge instructions.
Time Frame: Upon completion of surgery approximately 24 days post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of eligible patients
Groups:
- Activity Restriction: Discharge orders for activity restriction Activity Restriction: Standard post-operative activity instructions (i.e., no bending, twisting, or lifting more than 10 lbs for 4 weeks, no return to work until cleared to do so).
- Activity as Tolerated: Discharge orders written for activity as tolerated Activity as Tolerated: Instructions advising activity as tolerated and return to work based on patient discretion
Arm/Group | Activity Restriction | Activity as Tolerated
Number analyzed (Participants) | 19 | 18
percentage of eligible patients | 89 [65 to 98] | 50 [29 to 71]

2. Primary Outcome: Percentage Eligible Patients Participating in Study
Description: Percentage of those identified as being eligible who were enrolled.
Time Frame: 1 day, during the recruitment period from October 23 2020 to August 7, 2021
Population: All patients who were identified as being eligible and invited to participate.
Measure: Number (95% Confidence Interval); unit: percentage of eligible patients
Groups:
- All Eligible Patients: All eligible patients approached to participate.
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 48
percentage of eligible patients | 77 [62 to 87]

ADVERSE EVENTS:
Time Frame: Duration of follow-up for adverse events ranged from 288 days for the first patient randomized to 31 days for the last patient randomized.
Description: Attending surgeon and clinical reports.
Arm/Group | Activity Restriction | Activity As Tolerated
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

LIMITATIONS AND CAVEATS:
Primary limitations of the trial include limited enrollment compared to the original goal of 60 randomized patients due in part to the limitations in elective surgery during the Covid-19 pandemic. By design, the study is pragmatic, and primarily intended to evaluated methodologies for embedding randomization in the electronic record system of a regional health care center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT04520009/Prot_SAP_000.pdf